CLINICAL TRIAL: NCT05033223
Title: Psycho-traumatic Consequences of the COVID-19 Health Crisis Among Professionals in Emergency Services and SAMU: Multicenter Cohort Study (COVid in EmeRgency PROfessionnals Long Term)
Brief Title: Psycho-traumatic Consequences of the COVID-19 Health Crisis Among Professionals in Emergency Services
Acronym: COVER PRO LT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Elisa Letellier, Psycho-traumatic consequences of the COVID-19 health crisis among professionals in emergency services and SAMU: multicenter cohort study (COVid in EmeRgency PROfessionnals Long Term), Hospices Civils de Lyon
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL21_0311
Record Dates: First submitted 2021-09-01; First posted 2021-09-02 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Post Traumatic Stress Disorder
Keywords: post traumatic stress disorder; PTSD; emergency services; COVID-19; burn-out
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; COVID-19; Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Follow-up (Other)
  Interventions: Other: PTSD evaluation of emergency room staff 9 and 12 months after the end of second lockdown in France during COvid-19 pandemic

INTERVENTIONS:
Other: PTSD evaluation of emergency room staff 9 and 12 months after the end of second lockdown in France during COvid-19 pandemic — PCL-5 autoquestionnaire to make the PTSD diagnosis

SUMMARY:
The COVID-19 outbreak has been categorized as a pandemic and declared an international public health emergency by WHO. In this context, an exceptional mobilization and a complete reorganization of the organization of the healthcare offer was put in place.The investigators will study the psychological consequences among emergency department (ED) / SAMU (Service d'Aide Médicale Urgente) professionals exposed during the COVID-19 pandemic to high psychological stress due to work overload, changes in practices and fears of contamination.They will evaluate at 9 and 12 months after the end of the second lockdown (July December 2020), post-traumatic stress disorder (PTSD), personal and professional stress, anxiety and depression, burn-out and consumption of anxiolytic products. This is a multi-center study and includes doctors, DE interns and nurses, other paramedics and medical regulatory assistants working in one of the ED or SAMU working during phase 3 of the COVID-19 pandemic. It should make it possible to know the psychological load of the months following the epidemic among health professionals who worked in emergencies during this period and to understand their risk of occurrence of PTSD. These elements are also essential to improve the management of health crises and to put in place preventive measures for health professionals, in particular in anticipation of recurrences, second wave or future new episode.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Administrative and technical medical staff of the Hospices Civils de Lyon
* Contractual or holder
* Having participated in the COVER PRO study
* Working in one of the HCL phase 3 departments of the COVID-19 pandemic.
* Affiliated with a social security system
* Having signed an informed consent

Exclusion Criteria:

* Refusal to participate
* Major under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-01-16 (Actual); Study Completion 2022-01-16 (Actual)

PRIMARY OUTCOMES:
Existence of a Post Traumatic Stress Disorder (PTSD) at 12 months using PTSD Scale | 12 months after the end of the second Lockdown (December 2020)
  : Existence of a PTSD after the end of the second lockdown using the PCL-5 scale (Post Traumatic Stress Disorder Checklist, 20 items, self-questionnaire) validated in French for PTSD screening. The presence of a "probable PTSD" will be defined by a cut-off score of 31/80 and at least a positive response to one of the four questions asking if the symptoms were causing difficulties in relations with family, friends, work or in daily life

SECONDARY OUTCOMES:
Existence of a Post Ttraumatic Stress Disorder (PTSD) 9 months using PTSD Scale | 9months after the end of the second Lockdown (December 2020)
  Existence of a PTSD after the end of the second lockdown using the PCL-5 scale (Post Traumatic Stress Disorder Checklist, 20 items, self-questionnaire) validated in French for PTSD screening. The presence of a "probable PTSD" will be defined by a cut-off score of 31/80 and at least a positive response to one of the four questions asking if the symptoms were causing difficulties in relations with family, friends, work or in daily life
Anxiety evaluation at 12 months using HAD scale | 12months after the end of the second Lockdown (December 2020)
  Existence of anxious symptomatology assessed by the HAD scale. 14 items, cut-off score: 8 suspected disorder, 11: proven disorder
Anxiety evaluation at 9 months using HAD scale | 9months after the end of the second Lockdown (December 2020)
  Existence of anxious symptomatology assessed by the HAD scale. 14 items, cut-off score: 8 suspected disorder, 11: proven disorder
Depression evaluation at 12 months using HAD scale | 12months after the end of the second Lockdown (December 2020)
  Existence of depression symptomatology assessed by the HAD scale. 14 items, cut-off score: 8 suspected disorder, 11: proven disorder
Depression evaluation at 9 months using HAD scale | 9months after the end of the second Lockdown (December 2020)
  Existence of depression symptomatology assessed by the HAD scale. 14 items, cut-off score: 8 suspected disorder, 11: proven disorder
Presence of a Burn out at 12 months using the Maslach Burnot Inventory (MBI) scale | 12months after the end of the second Lockdown (December 2020)
  Burnout characterized by the Maslach burnout inventory scale. All MBI items are scored using a 7 level frequency ratings from "never" to "daily." The MBI has three component scales: emotional exhaustion (9 items), depersonalization (5 items) and personal achievement (8 items). Each scale measures its own unique dimension of burnout.
Presence of a Burn out at 9 months using the MBI scale | 9months after the end of the second Lockdown (December 2020)
  Burnout characterized by the Maslach burnout inventory scale. All MBI items are scored using a 7 level frequency ratings from "never" to "daily." The MBI has three component scales: emotional exhaustion (9 items), depersonalization (5 items) and personal achievement (8 items). Each scale measures its own unique dimension of burnout.
Work-related stress measured using Karasek questionnaire at 12 months | 12months after the end of the second Lockdown (December 2020)
  Work-related stress measured using Karasek questionnaire at 12 months
Work-related stress measured using Karasek questionnaire at 9 months | 9months after the end of the second Lockdown (December 2020)
  Work-related stress measured using Karasek questionnaire at 9 months
Consumption of psychoactive substances at 12 months | 12months after the end of the second Lockdown (December 2020)
  Change in the consumption of psychoactive substances at 12 months
Percentage of patients with psychological Support at 12 months | 12months after the end of the second Lockdown (December 2020)
  Percentage of patients who benefit from a psychological support at 12 months
Mean number of days of sick leave at 12 months | 12months after the end of the second Lockdown (December 2020)
  Mean number of days of sick leave at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Accueil des Urgences, Pierre-Bénite, France